CLINICAL TRIAL: NCT05286424
Title: Lipofilling: Optimal Harvesting Techniques for Breast Reconstruction After Mastectomy in Plastic Aesthetic and Reconstructive Surgery - a Pilot Study
Brief Title: Lipofilling: Optimal Harvesting Techniques for Breast Reconstruction After Mastectomy in Plastic Aesthetic and Reconstructive Surgery
Acronym: LipoTech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Joanneum Research Forschungsgesellschaft mbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 32-487 ex 19/20
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: The Impact of Adipose Tissue Quality on Fat Graft Retention
Keywords: fat graft, adipose tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: fat grafting — Fat will be removed from abdomen or legs, processed and re-injected into grafting sites.
  Other Names: lipofilling

SUMMARY:
The primary aim of this project is to standardize the method for lipofilling by identifying the best technique. In this context, the study will investigate the impact of adipose tissue composition and ideal quantity of the injected fat particularly in view of resorption rate. Correlations between adipose tissue composition, amount of transferred fat, already existing subcutaneous fat layer at the grafting site and resorption rate will be made.

The punch biopsy and the non-invasive Lipometer measurements to determine the subcutaneous fat layer thickness in the harvesting and grafting region will be performed in 10 female subjects that undergo elective lipofilling.

The study was registered on Clinicaltrials.gov after start of recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Women, age 18-70 years (limited upwards due to the indication for lipofilling and the amount of possible secondary diseases)
* History of BRCA1 and BRCA2 - positive breast cancer with following subcutaneous mastectomy
* Planned, elective breast-lipofilling
* Thickness of the skin and subcutaneous fat layer of min. 1 cm (detected via sonography)
* Currently healthy individual, willing to participate in this study

Exclusion Criteria:

* Previous surgery at the harvesting site (e.g. caesarian section)
* Pregnancy or planned pregnancy
* Current or preceded chemotherapy
* Preceded radiatio
* Unable to fully understand study procedures and to provide informed consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Fat grafting after mastecomy is studied, therefore a gender bias is not avoidable.
Enrollment: 10 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Adipose tissue dependent take rate | 12-24 months
  Detect an adipose tissue composition-dependent take rate

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Universität Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided